CLINICAL TRIAL: NCT04133558
Title: Association of Lung Microbiota With Intensive Care Unit Mortality in ARDS Patients: MicrA Study
Brief Title: Pulmonary Microbiota and ARDS Mortality
Acronym: MicrA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bordeaux (Other)
Responsible Party: Principal Investigator, Dr Pauline Esteves, Doctor, University of Bordeaux
Other Study IDs: MicrA
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: acute respiratory distress syndrome; microbiota; intensive care unit
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tracheal aspirate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: tracheal aspirate during routine care — tracheal aspirate during routine care

SUMMARY:
Acute respiratory distress syndrome (ARDS) is due to diffuse and severe lung inflammation. Despite intensive research, few therapeutics have emerged and treatment is still mostly symptomatic. As lung microbiota seems to be associated with lung inflammation in numerous chronic respiratory diseases, this study aims to analyse the correlation between lung microbiota and mortality.

DETAILED DESCRIPTION:
ARDS is caused by diffuse intense lun inflammation. Its mortality rate is still about 40%. Despite decades of research, few therapeutics have emerged. Treatment is based on the treatment of ARDS cause, if possible and on protective ventilation, curare use and prone position. For more severe cases, nitric monoxide inhalation and extra-corporeal membrane oxygenation can be considered. Nevertheless, no treatment specifically addresses lung inflammation. Lung microbiota has been shown to be associated with lung inflammation in asthma, chronic obstructive disease and cystic fibrosis. Lung microbiota also plays a role in lung immunity. Regarding specifically ARDS, one study correlated lung microbiota with the occurrence of non-infectious ARDS in trauma patients. Thi study therefore aims to analyse the correlation between lung microbiota at admission to ICU for ARDS with mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 year-old admitted to intensive care unit
* ARDS according to Berlin criteria
* Needing oro-tracheal intubation for mechanical ventilation
* Within the first 48 hours of ARDS evolution

Exclusion Criteria:

* Guardianship or curatorship
* Prisoners
* No health insurance
* No legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS patients needing oro-tracheal intubation for mechanical ventilation in ICU
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
lung bacteriobiota and ICU mortality | at admission
  Comparison of lung bacteriobiota alpha diversity between ARDS ICU survivors and non-survivors

SECONDARY OUTCOMES:
lung mycobiota and ICU mortality | at admission
  Comparison of lung mycobiota alpha diversity between ARDS ICU survivors and non-survivors
lung mycobiota and 1-month mortality | microbiota : at admission, mortality: 1 month after inclusion
  Comparison of lung mycobiota alpha diversity between ARDS 1-month survivors and non-survivors
lung bacteriobiota and ICU mortality | at admission
  Analysis of lung bacteriobiota beta diversity between ARDS ICU survivors and non-survivors
lung bacteriobiota and 1-month mortality | microbiota : at admission, mortality: 1 month after inclusion
  Analysis of lung bacteriobiota beta diversity between ARDS 1-month survivors and non-survivors
lung mycobiota and ICU mortality | at admission
  Analysis of lung mycobiota beta diversity between ARDS ICU survivors and non-survivors
lung mycobiota and 1-month mortality | microbiota : at admission, mortality: 1 month after inclusion
  Analysis of lung mycobiota beta diversity between ARDS 1-month survivors and non-survivors
bacteria and ICU mortality | at admission
  Association of bacteria with ARDS ICU mortality by LefSe method
bacteria and 1-month mortality | microbiota : at admission, mortality: 1 month after inclusion
  Association of bacteria with ARDS 1-month mortality by LefSe method
fungi and ICU mortality | at admission
  Association of fungi with ARDS ICU mortality by LefSe method
fungi and 1-month mortality | microbiota : at admission, mortality: 1 month after inclusion
  Association of fungi with ARDS 1-month mortality by LefSe method

CONTACTS AND LOCATIONS:
Locations (1):
- Medical intensive care unit, Pellegrin hospital, Bordeaux, Nouvelle-Aquitaine, France

IPD SHARING:
Plan to Share IPD: No